CLINICAL TRIAL: NCT04322591
Title: Chemotherapy or Chemotherapy Plus PD-1 Antibody in RET Fusion Positive Advanced Non-small Cell Lung Cancer ( Poseidon Study）
Brief Title: Chemotherapy or Chemotherapy Plus PD-1 Antibody in RET Fusion Positive Advanced NSCLC Patitnts: the POSEIDON Trial
Acronym: POSEIDON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, professor, Hunan Province Tumor Hospital
Other Study IDs: POSEIDON
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: PD-L1 ;RET Fusion Lung Cancer Patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the efficacy and safety of chemotherapy or chemotherapy plus PD-1 antibody in RET Fusion Positive Advanced Non-small Cell Lung Cancer.

DETAILED DESCRIPTION:
This study aims to explore the efficacy and safety of chemotherapy or chemotherapy plus the PD-1 antibody in RET Fusion Positive Advanced Non-small Cell Lung Cancer. We aim to enrolled 100 patients in this study, the primary endpoint was PFS.

ELIGIBILITY:
Inclusion Criteria:

* ≥18，Advanced Non-squamous Non-small Cell Lung Cancer Confirmed by Histopathology
* RET Fusion Positive
* First Diagnosis and Treatment
* Treatment Plan is Chemotherapy or Chemotherapy plus PD-1 antibody

Exclusion Criteria:

* - Patients received antitumor treatment before
* Patients with contraindication of chemotherapy
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RET Fusion Positive Advanced Non-squamous Non-small Cell Lung Cancer Confirmed by NGS
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2025-03-24 (Estimated)

PRIMARY OUTCOMES:
PFS | may 2020- may 2021 (1 year)
  Progression free survival time

SECONDARY OUTCOMES:
ORR | may 2020- may 2021 (1 year)
  Overal response rate
OS | may 2020- may 2021 (1 year)
  Overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China